CLINICAL TRIAL: NCT06777199
Title: A Comparative Study to Assess the Role of Selective Dorsal Neurectomy Versus Pulsed Radiofrequency Neuromodulation Versus Intraglanular Hyaluronic Acid Injection for Patients With Lifelong Premature Ejaculation: a Randomized Clinical Trial
Brief Title: A Comparative Study of Selective Dorsal Neurectomy, Pulsed Radiofrequency Neuromodulation, and Intragranular Hyaluronic Acid Injection for Premature Ejaculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Hamdy Ahmed (Other)
Responsible Party: Sponsor-Investigator, Ahmed Hamdy Ahmed, Urology Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-273-2022
Record Dates: First submitted 2024-12-20; First posted 2025-01-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Premature Ejaculation
Keywords: lifelong premature ejaculation; Microscopic Selective Dorsal Neurectomy; intraglanular Hyaluronic acid; pulsed radiofrequency ablation
MeSH Terms: conditions — Premature Ejaculation | interventions — Prolactin-Releasing Hormone; Injections

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group design with three independent intervention arms. Thirty male patients with lifelong premature ejaculation (PE) were randomly assigned into one of the following treatment groups:
  Group A: Selective dorsal neurectomy performed under spinal anesthesia. Group B: Pulsed radiofrequency nerve ablation under local anesthesia. Group C: Intraglanular hyaluronic acid injection under local anesthesia. Participants remain in their respective groups throughout the study, and outcomes, including intravaginal ejaculatory latency time (IELT), Arabic Index of Premature Ejaculation (AIPE), and Premature Ejaculation Diagnostic Tool (PEDT) scores, are evaluated at 1 month and 3 months post-intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microscopic Selective Dorsal Neurectomy Group (Experimental): Participants in this group will undergo microscopic selective dorsal neurectomy (SDN). The procedure involves partial transection of the dorsal penile nerves under spinal or local anesthesia to reduce sensitivity of the glans penis. Post-procedure, outcomes will be assessed at 1 and 3 months using stopwatch-measured intravaginal ejaculatory latency time (IELT) and validated questionnaires (AIPE, PEDT, and PEP).
  Interventions: Procedure: Microscopic Selective Dorsal Neurectomy (SDN)
- Pulsed Radiofrequency Nerve Ablation Group (Experimental): Participants in this group will receive pulsed radiofrequency (PRF) neuromodulation targeting the dorsal penile nerves. The procedure involves delivering low-energy radiofrequency pulses through an RF cannula inserted into the flaccid penile skin. The goal is to reduce glans sensitivity and improve IELT. Outcomes will be evaluated at 1 and 3 months using stopwatch-measured IELT and validated questionnaires (AIPE, PEDT, and PEP).
  Interventions: Procedure: Pulsed Radiofrequency (PRF) Nerve Ablation
- Intraglanular Hyaluronic Acid Injection Group (Experimental): Participants in this group will receive intraglanular hyaluronic acid (HA) injections. The circumference of the glans penis will be divided into multiple sections, and HA gel will be injected under local anesthesia to reduce glans sensitivity. Outcomes will be assessed at 1 and 3 months using stopwatch-measured IELT and validated questionnaires (AIPE, PEDT, and PEP).
  Interventions: Procedure: Intraglanular Hyaluronic Acid (HA) Injection

INTERVENTIONS:
Procedure: Microscopic Selective Dorsal Neurectomy (SDN) — Selective dorsal neurectomy (SDN) involves microsurgical dissection and partial transection of the dorsal penile nerves to reduce glans sensitivity.
  The procedure is performed under spinal anesthesia or local anesthesia with 1% lidocaine.
  A midline or dorsal sub-coronal incision is made 1 cm proximal to the coronal sulcus.
  The skin is retracted, exposing the Dartos fascia and Buck's fascia to reach the neurovascular bundle (two dorsal penile nerves lateral to two dorsal penile arteries).
  Every other nerve on either side of the corpora cavernosa is transected to damage approximately 50% of the nerve supply to the glans.
  Suturing is done using 7-0 or 8-0 prolene sutures, and the incision is closed. Patients are evaluated at 1 month and 3 months post-procedure for IELT, AIPE, and PEDT scores to determine success.
  Arms: Microscopic Selective Dorsal Neurectomy Group
Procedure: Pulsed Radiofrequency (PRF) Nerve Ablation — Pulsed radiofrequency (PRF) nerve ablation aims to reduce sensitivity of the dorsal penile nerves using low-energy radiofrequency pulses.
  Under sterile conditions, a 22-gauge RF cannula (5-cm-long, 10-mm active tip) is inserted into the flaccid penile skin at the 1-o'clock position for the right dorsal penile nerve.
  Sensory stimulation testing is performed at 50 Hz to identify the point of maximum glans sensitivity.
  Pulsed radiofrequency is applied at an energy output of 45 V for 180 seconds at 42°C (using the NeuroTherm generator).
  The procedure is repeated at the 11-o'clock position for the left dorsal penile nerve, ensuring both sides are treated.
  The goal is to ablate sensation over as large an area of the glans as possible without causing permanent nerve damage.
  Post-procedure, patients are evaluated at 1 and 3 months for IELT, AIPE, and PEDT scores.
  Arms: Pulsed Radiofrequency Nerve Ablation Group
Procedure: Intraglanular Hyaluronic Acid (HA) Injection — Intraglanular hyaluronic acid (HA) injection involves administering HA gel into the glans penis to reduce its sensitivity.
  The circumference of the glans penis is divided into three circles (1 cm apart, starting from the base), and each circle is further divided into quarter circles.
  Topical anesthetic cream (Emla®, lidocaine 25 mg + prilocaine 25 mg) is applied for 30 minutes to numb the glans.
  Using two prefilled syringes of HA gel (Hyabell Ultra® 24 mg/ml with 0.3% lidocaine), 12 injections are administered into the deep dermis of the glans using a 27-G needle.
  Each injection site receives 0.25 ml of HA gel following the multiple puncture technique.
  Patients are evaluated at 1 and 3 months for IELT, AIPE, and PEDT scores to assess efficacy.
  Arms: Intraglanular Hyaluronic Acid Injection Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of three treatment methods for lifelong premature ejaculation (PE) in adult males. The main questions this study aims to answer are:

Does selective dorsal neurectomy, pulsed radiofrequency nerve ablation, or hyaluronic acid injection prolong intravaginal ejaculatory latency time (IELT)? What are the differences in patient satisfaction and safety among the three treatments?

In this study:

Participants will be randomized into three groups (10 patients each). Group 1 will undergo selective dorsal neurectomy under local or spinal anesthesia.

Group 2 will receive pulsed radiofrequency nerve ablation sessions. Group 3 will have hyaluronic acid injections into the glans penis under local anesthesia.

Researchers will measure treatment outcomes using:

Stopwatch measurements of IELT. Patient-reported questionnaires (IPE, PEP). International Index of Erectile Function-5 (IIEF-5) to confirm no erectile dysfunction.

DETAILED DESCRIPTION:
This randomized clinical trial aims to assess the efficacy and safety of three treatment modalities for lifelong premature ejaculation (PE) in adult males. Premature ejaculation is a common male sexual dysfunction that significantly impacts quality of life, affecting relationships and psychological well-being. The study will compare three therapeutic approaches: selective dorsal neurectomy, pulsed radiofrequency nerve ablation, and intraglanular hyaluronic acid injection.

Study Population:

Male patients aged 18 years and older. Participants must have lifelong PE that has not responded to or cannot be continued with medical treatment.

Patients with erectile dysfunction, severe comorbidities, or recent use of SSRIs or topical anesthetics will be excluded.

Intervention Groups:

Selective Dorsal Neurectomy (SDN):

Performed under spinal or local anesthesia. Involves microsurgical dissection of the dorsal penile nerves to reduce glans sensitivity.

Pulsed Radiofrequency Nerve Ablation (PRF):

Involves neuromodulation of the dorsal penile nerves using pulsed radiofrequency energy.

The goal is to reduce glans sensation while preserving nerve function.

Hyaluronic Acid Injection:

Hyaluronic acid is injected into the glans penis using the multiple puncture technique under local anesthesia to reduce sensitivity.

Outcome Measures:

Primary Outcomes:

Prolongation of intravaginal ejaculatory latency time (IELT) using stopwatch measurements.

Improvement in patient-reported outcomes via validated questionnaires (IPE, PEP).

Secondary Outcomes:

Improvement in patient and partner sexual satisfaction. Presence of voluntary control of ejaculation. Reduction in stress and psychological distress.

Study Design:

A total of 30 patients will be randomized into three equal groups (10 patients per group).

The follow-up period includes evaluations at 1 month and 3 months post-intervention.

Diagnostic tools include IELT stopwatch measures, penile duplex ultrasound, and questionnaires.

Statistical Analysis:

Data will be analyzed using SPSS software. Descriptive statistics (mean, standard deviation) and comparative tests (paired t-tests, Chi-square tests) will determine the significance of results.

This study aims to provide evidence-based guidance on the optimal treatment strategy for lifelong premature ejaculation, focusing on efficacy, safety, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* all male patients ≥ 18 years old who are having regular sexual life and suffering from lifelong premature ejaculation, not responding to medical treatment or not willing to continue on medical treatment

Exclusion Criteria:

* Patients suffering from ED
* Patients suffering of several debilitating co-morbidities (uncontrolled DM, on corticosteroids or receiving immunosuppression therapy)
* Patients suffering of neurological disorders
* Patients receiving any kind of SSRIs or topical anesthetics within 3 months to treat LPE
* Patients suffering from any other form of PE (i.e. acquired, subjective, variable PE)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Prolongation of intravaginal ejaculatory latency time (IELT) | 1 month and 3 months
Improvement in patient-reported outcomes using the Index of Premature Ejaculation (IPE) questionnaire | 1 month and 3 months
  The IPE questionnaires scoring is normally classified to measure severity as follows:
  • IPE scoring (the lower the score, the higher the PE severity): Severe PE: 7-13 Moderate PE: 14-19 Mild to Moderate PE: 20-25 Mild PE: 26-30 No PE: 31-35
Improvement in patient-reported outcomes using the Premature Ejaculation Diagnostic Tool (PEDT) questionnaire | 1 month and 3 months
  The PEDT questionnaire scoring is normally classified to measure severity as follows:
  • PEDT scoring (the lower the score, the lower the PE probability): Highly PE: ≥11 Borderline PE: 9-10 No PE: ≤ 8

SECONDARY OUTCOMES:
Improvement in patient and partner sexual satisfaction | 1 month and 3 months
  Sexual Satisfaction Scale (SSS)
  Minimum Value: 4 (very dissatisfied across all items) Maximum Value: 20 (very satisfied across all items)
  Scoring: The SSS evaluates sexual satisfaction using four items rated on a 5-point scale:
  1 = Very dissatisfied 2 = Dissatisfied 3 = Neutral 4 = Satisfied 5 = Very satisfied
  Interpretation: Higher scores indicate greater overall sexual satisfaction for the patient and their partner.
  Assessment Method:
  Patients and their partners independently complete the Sexual Satisfaction Scale (SSS) questionnaire.
  The total score is calculated separately for the patient and partner. The average score across both individuals is used for reporting overall satisfaction.
Presence of voluntary control of ejaculation | 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Faculty of Medicine, Giza, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided